CLINICAL TRIAL: NCT05104060
Title: The Effects of Manual Therapy and Scapular Exercise for the Pectoralis Minor in Individuals With Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Cheng-Hsin General Hospital (Other)
Responsible Party: Principal Investigator, Yin-Liang Lin, Assistant Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM110136E
Record Dates: First submitted 2021-09-28; First posted 2021-11-02 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Shoulder Pain; Shoulder Impingement; Scapular Dyskinesis
Keywords: pectoralis minor length; pectoralis minor index; scapular kinematic
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pectoralis minor intervention group (Experimental): The participants in pectoralis minor group will received manual therapy for pectoralis minor by investigators, the technique including stretch and soft tissue mobilization. The participants asked to perform the scapular control exercise and shoulder strength exercise. Participants will be correct scapular resting position and then do elevation in scapular plane.Four exercises for shoulder strength will do shoulder flexion, abduction, internal and external rotation with thera-band.
  Interventions: Procedure: pectoralis minor intervention group
- shoulder strengthening group (Active Comparator): The participants in the scapular strengthening group will be asked to do four exercises for shoulder strength, including shoulder flexion, abduction, internal and external rotation with thera-band.
  Interventions: Procedure: shoulder strengthening group
- Healthy subject group (No Intervention): Healthy participants will be recruited. No Intervention will be provided. The correlation between measures of pectoralis minor length and scapular kinematics will be assessed. Measurement will be the same as pectoralis minor intervention group and shoulder strengthening group

INTERVENTIONS:
Procedure: pectoralis minor intervention group — The subjects in pectoralis minor group will received manual therapy for pectoralis minor by physical therapist, the technique including stretch and soft tissue mobilization. The subjects asked to perform the scapular control exercise and shoulder strength exercise.Subjects will be correct scapular resting position and then do elevation in scapular plane.Four exercises for shoulder strength will do shoulder flexion, abduction, internal and external rotation with thera-band.
  Arms: pectoralis minor intervention group
Procedure: shoulder strengthening group — The subjects in the scapular strengthening group will be asked to do four exercises for shoulder strength, including shoulder flexion, abduction, internal and external rotation with thera-band.
  Arms: shoulder strengthening group

SUMMARY:
Shoulder pain is the third common problem, after problems of spine. Abnormal scapular kinematics, so called scapular dyskinesis, is believed to be associated with shoulder pain. Studies showed that individuals with shoulder problems demonstrate less upward rotation, posterior tilt and external rotation during shoulder movement. The shortness of the pectoralis minor (PM) is one of the factors leading to scapular dyskinesis. Short pectoralis minor has been shown to prevent scapula from tilting posterior and rotating externally during shoulder motion. The decreased scapular posterior tilt and external rotation may decrease subacromial space and result in impingement. However, although many assessment methods have been used to assess PM tightness or shortness, no study has tested the validity of these testing methods. Moreover, although stretching exercises for PM have been shown to increase the PM length, previous studies found that PM stretching exercises did not restore scapular kinematics and did not further decrease pain and improve function. Shoulder pain and discomfort has also been reported during stretching. Therefore, rather than stretching exercise, other types of treatment that can specifically increase the PM length and restore scapular kinematics may be needed. Manual therapy could specifically increase the flexibility of PM, and scapular orientation exercises could improve scapular kinematics. These types of treatment may be better options. However, to our knowledge, no study has investigated whether manual therapy combined with scapular orientation exercises could improve scapular kinematics, pain and function. Therefore, the first part of this study is to investigate which tests for length or tightness of PM can predict the scapular dyskinesis. The second part of the study is to investigate the effects of manual therapy and scapular orientation training on PM length, scapular kinematics, pain, and function in subjects with shoulder pain. In the first part of the study, 67 healthy subjects will be recruited. In the second part, 62 patients with shoulder pain will be recruited and randomized into either a PM treatment group or a control group. While no treatment will be provided for the healthy subjects in the first part, subjects with shoulder pain in the second part will receive 12 sessions of treatment in 4-6weeks, with 30-40 minutes per session. Patients in the control group will receive general shoulder strengthening exercise, while patients in the PM treatment group will have additional manual therapy and scapular orientation exercise. The measures include tests of PM length, scapular kinematics in the first and second parts, and pain and shoulder disability were also additionally assessed in the second part.

ELIGIBILITY:
Inclusion Criteria(patients with shoulder pain) :

1. the patients with shoulder pain from 20 - 60 years old
2. Active arm elevation close to 150 degrees
3. Shoulder pain at least 3 months

Inclusion Criteria (healthy people) :

1. the people from 20 - 40 years old
2. no any symptoms or injuries on shoulder one year ago

Exclusion Criteria:

1. Adhesive capsulitis
2. Pathologies of cervical origin
3. History of acute trauma, previous surgery, or fracture in the affected shoulder
4. Corticoid injection in the last 3 months
5. Platelet Rich Plasma injection in the last 1 year
6. Other manual and exercise physical therapy in the last 6 weeks
7. Anyone suffering from neurological diseases and nerve damage
8. Vulnerable subjects

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Pectoralis minor length | Change from baseline pectoralis minor length after 12 times intervention up to 6 weeks
  Measurement of pectoralis minor length: distance between coracoid process and fourth rib taken with a tape measure on resting position.
Pectoralis minor index | Change from baseline pectoralis minor index after 12 times intervention up to 6 weeks
  The pectoralis minor length was divided by the participant's height and multiplied by 100 to calculate the pectoralis minor index
Pectoralis minor tightness test I | Change from baseline pectoralis minor tightness test I after 12 times intervention up to 6 weeks
  Pressed the coracoid process of the subjects to make the scapula flat on the treatment bed.If flat the bed for negative,unable to flat the bed for positive.
Pectoralis minor tightness test II | Change from baseline pectoralis minor tightness test II after 12 times intervention up to 6 weeks
  Subjects will forward flexion 30 degrees,and pressed the coracoid process.If physical therapist felt tightness for positive.
Round shoulder posture test I | Change from baseline round shoulder posture test I after 12 times intervention up to 6 weeks
  Measured the distance between the posterior border of the acromion and the table surface.
Round shoulder posture test II | Change from baseline round shoulder posture test II after 12 times intervention up to 6 weeks
  Measured the vertical distance between the posterior acromion and the treatment bed,then divided by thorax thickness and multiplied by 100.
Scapular kinematics | Change from baseline scapular kinematics after 12 times intervention up to 6 weeks
  Scapular kinematics, including anterior/posterior tilt, upward/downward rotation, and internal/external rotation in scapula plan elevation at 30°, 60°, 90°, and 120°, will be calculated and will be described with degree (°).

SECONDARY OUTCOMES:
Visual analog scale | Change from baseline visual analog scale after 12 times intervention up to 6 weeks
  Scores ranging from 0 (no pain) to 10 (maximum pain)
Disabilities of the Arm, Shoulder, and Hand (DASH) | Change from baseline DASH after 12 times intervention up to 6 weeks
  A maximum score of 100 indicates the worst possible condition
Patient-Specific Functional Scale (PSFS) | Change from baseline PSFS after 12 times intervention up to 6 weeks
  Identify 3 important activities that they were unable to perform. A minimum score of 0 is unable to engage in these activities, and a maximum score of 10 can still perform these activities as efficiently as before without shoulder pain.
Global rating of change (GRC) | After 12 times intervention up to 6 weeks
  Independently score self-perceived improvement in a patient. A minimum score of -5 is the worse situation compared to before treatment. Compared to before treatment, a score of 0 means no change.Compared to before treatment, a score of 5 means full recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Liang Lin, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (2):
- Taiwan (2):
  - National Yang-Ming University, Taipei
  - Cheng Hsin General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No